CLINICAL TRIAL: NCT03142412
Title: Lupus Interval Monitoring to Manage Disease Flare and Enable Treatment Optimization
Acronym: LIFT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: DxTerity Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: DXT-MCD-AD01-LIFT
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Systemic Lupus Erythematosus; Lupus; Lupus Erythematosus; Lupus Erythematosus, Systemic
Keywords: Lupus; SLE; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop a test to characterize and monitor SLE disease activity status from a participant's home by analyzing the gene expression from participant self-collected blood samples using a novel fingerstick collection kit.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE or lupus) is a chronic inflammatory autoimmune disorder of poorly understood etiology associated with a wide range of symptoms and physical findings.

Many patients have incompletely controlled disease progressing to end-stage organ involvement. Recognizing and predicting flares and under associated organ damage would facilitate better treatment timing and selection. Recent improvements in care have dramatically enhanced the survival of lupus patients but increased mortality remains a major concern and current treatments for lupus remain inadequate. Development of novel therapies to manage lupus has been hampered by several challenges, including poorly understood pathogenesis, the heterogeneity of disease activity across and within patient populations, and difficulties conducting interventional studies. There remains a need for reliable and timely monitoring of disease activity and degree of organ damage to adequately evaluate response to treatments and long-term outcome. It is also important to differentiate genuine lupus activity and flares from another intercurrent disease such as infection.

To fill this gap, panels of reliable biomarkers that can classify patients with lupus into more homogenous subsets that are linked to disease activity are needed. Such a panel can be developed from signatures found in lupus patients' transcriptome sequencing data. DxTerity's proprietary DxCollect® Microcollector Device (MCD) is intended to facilitate the collection, stabilization, and shipping of a microsample (about 150μL) of blood. This microsample provides sufficient amounts of quality RNA to perform transcriptome sequencing, allowing identification and validation of candidate biomarker signatures. A rapid blood test to monitor and predict disease activity and treatment response would be an innovative diagnostic product. It could bring significant clinical benefits by enabling the individualized lupus monitoring and treatment to better control the disease and slow organ damage. This may assist with unburdening healthcare costs, help identify flares before they happen, and dramatically improve the management of lupus.

The study will collect participant self-collected blood samples from a fingerstick collection kit that can be done from home and self-reported information from up to 2500 participants for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18 or older
2. Have a permanent address in the United States for the duration of the study
3. Have an email address and access to the internet for the duration of the study
4. Able to provide informed consent
5. Self-reported diagnosis of lupus

Exclusion Criteria:

1. None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with Systemic Lupus Erythematosus (SLE).
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2017-04-17 (Actual); Primary Completion 2021-10-17 (Estimated); Study Completion 2021-10-17 (Estimated)

PRIMARY OUTCOMES:
Obtain blood samples and associated clinical and demographic data from participants diagnosed with Systemic Lupus Erythematosus (SLE) | 4.5 years
  Obtain blood samples and associated clinical and demographic data from participants diagnosed with Systemic Lupus Erythematosus (SLE) to develop a blood test to characterize SLE status by analyzing gene expression from blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- DxTerity Diagnostics, Compton, California, United States

IPD SHARING:
Plan to Share IPD: No